CLINICAL TRIAL: NCT04693221
Title: Optimization of the Parameters of Vagal Nerve Stimulation in Pharmaco- Resistant Epileptic Patients Based on a Surface EEG Index of Functional Connectivity (PLI: Phase Lag Index): a Randomized Double-blind Multicenter Controlled Study.
Brief Title: Optimization of the Parameters of Vagal Nerve Stimulation
Acronym: OPSTIMVAG
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-05; 2020-A02657-32 (Other: ID-RCB)
Record Dates: First submitted 2020-12-31; First posted 2021-01-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Epilepsy
Keywords: epilepsy; vagal nerve stimulation; phase lag index
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Sham Comparator): VNS therapy with randomly-set combination of parameters (similar to current practice)
  Interventions: Other: EEG
- Experimental (Experimental): VNS therapy with set combination of parameters chosen based on the lowest phase lag index
  Interventions: Other: Choice of VNS set of parameters based on the lowest PLI; Other: EEG

INTERVENTIONS:
Other: Choice of VNS set of parameters based on the lowest PLI — Vagal nerve stimulation according to PLI results.
  Arms: Experimental
Other: EEG — Patient will have an EEG and 12 sets of parameters will be tested. EEG results will be analyzed which will allow to determine the set involving the lowest phase lag index.

SUMMARY:
Vagal nerve stimulation (VNS) is one of the neuromodulation techniques that can be indicated in patients suffering from refractory epilepsies, especially when an open resection has failed or is not indicated. However to date it is not possible to predict which patients will respond and what are the best parameters of stimulation to be set (pulse width, frequency and intensity). It has been shown that responders to VNS have reduced interictal cortical synchronicity on scalp EEG based on phase lag index (PLI), a marker of functional connectivity (Fc) The aim of this study is to test the following hypothesis: setting the parameters of stimulation on the basis of the lowest values of Phase Lag Index (PLI) obtained on scalp EEG with different settings of parameters (as compared with a randomly chosen set of commonly used parameters) will increase the rate of responders to VNS.

ELIGIBILITY:
Inclusion Criteria:

* Male or female epileptic patients over 12 years of age
* Suffering from pharmaco-resistant epilepsy
* With newly implanted VNS Aspire SR device
* Surgery performed in the previous 6 months
* Electrode impedance should be within normal range ( < 4000 Ohms)
* Auto-stim mode working properly
* Mean number of seizures of at least (average 4 (mean value) / months during the baseline period)
* Patient, parents or legally representatives who have given written informed consent to allow the study data collection and procedures

Exclusion Criteria:

* Difficulty to read or understand the French language, or inability to understand the information regarding the study
* Total patient's IQ below 64
* Subject in exclusion period due to enrolment in another study
* Patient with postoperative left vocal cord paralysis
* Patient on VNS since more than 6 months

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2026-12-12 (Estimated)

PRIMARY OUTCOMES:
Mean number of seizures per month | Change from baseline to 6 months
Mean number of seizures per month | Change from baseline to 12 months

SECONDARY OUTCOMES:
Number of responders in each group | Change from baseline to 6 months
Number of responders in each group | Change from baseline to 12 months
Number of generalized seizures | Change from baseline to 6 months
Number of generalized seizures | Change from baseline to 12 months
Number of seizures with falls | Change from baseline to 6 months
Number of seizures with falls | Change from baseline to 12 months
Number of seizures with alteration of consciousness | Change from baseline to 6 months
Number of seizures with alteration of consciousness | Change from baseline to 12 months
Score of depression | Change from baseline to 6 months
  NDDI-E
Score of depression | Change from baseline to 12 months
  NDDI-E
Score of anxiety | Change from baseline to 6 months
  GAD-7
Score of anxiety | Change from baseline to 12 months
  GAD-7
Score of quality of life | Change from baseline to 6 months
  QUOLIE 31
Score of quality of life | Change from baseline to 12 months
  QUOLIE 31

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (18):
- France (18):
  - Department of functional explorations of the nervous system, CHU, Amiens, France
  - Neuropediatrics department, CHU Angers, Angers, France
  - Neurology Department, CHU Bordeaux, Bordeaux, France
  - Clinical neurophysiology, CHU Dijon, Dijon, France
  - Epilepsy neurophysiopathology department, CHU Grenoble, Grenoble, France
  - Clinical neurophysiology, CHU Lille, Lille, France
  - HCL Lyon, Lyon, France
  - Department of clinical neurophysiology, Hôpital La Timone, APHM, Marseille, France
  - Neurosurgery Department, CHRU Nancy, Nancy, France
  - Neurosurgery Department, CHU Nantes, Nantes, France
  - Neurosurgery Department, APHP, Paris, France
  - Neurophysiology Department, Paris, France
  - Epileptology Department, CHU Rennes, Rennes, France
  - Neurophysiology Department, CHU Rouen, Rouen, France
  - Neurology Department, CHU Strasbourg, Strasbourg, France
  - Neurophysiological explorations, Hôpital Pierre Paul Riquet, Purpan, Toulouse, France
  - Neurology and clinical neurophysiology, CHU Bretonneau, Tours, France
  - Hôpital St Joseph St Luc, Lyon, FRA

IPD SHARING:
Plan to Share IPD: No